CLINICAL TRIAL: NCT04806763
Title: Myopia Control With Orthokeratology Contact Lenses in Spain
Acronym: MCOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menicon Co., Ltd. (Industry)
Collaborators: Universidad Europea de Madrid (Other); Aston University (Other); Clinica novovision (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCOS
Record Dates: First submitted 2021-03-10; First posted 2021-03-19 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Myopia, Progressive; Children, Only; Contact Lens Complication; Perception, Self; Axial Myopia
MeSH Terms: conditions — Myopia, Degenerative

STUDY DESIGN:
Intervention Model Description: Prospective, controlled, longitudinal
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Menicon Z Night (Experimental): The experimental group is allocated to wear Menicon Z Night orthokeratology contact lenses for two years
  Interventions: Device: Menicon Z Night
- Glasses (Active Comparator): The active comparator includes a group that was allocated to wear distance, single-vision glasses for two years
  Interventions: Device: Control

INTERVENTIONS:
Device: Menicon Z Night — To assess the use of Menicon Z Night contact lenses for reducing myopia progression in children
  Arms: Menicon Z Night
Device: Control — Distance, single-vision glasses were used as control
  Arms: Glasses

SUMMARY:
The purpose of this prospective study is to assess the efficacy, safety and patient-reported outcomes of the Menicon Z Night orthokeratolgy contact lens for reducing myopia progression in children.

DETAILED DESCRIPTION:
The purpose of this prospective study is to assess the efficacy, safety and patient-reported outcomes of the Menicon Z Night orthokeratolgy contact lens for reducing myopia progression in children in comparison with a group of distance, single-vision glasses over a 2-year period. Efficacy was evaluated by assessing differences in the axial length between groups. Safety was evaluated by comparing the incidence of adverse events between groups. Differences between groups in patient-reported outcomes were evaluated using a questionnaire that assessed vision-related quality-of-life measures.

ELIGIBILITY:
Inclusion Criteria:

* Be 6 to 12 years of age, both ages inclusive
* A low-to-moderate level of myopia (between -0.75 and -4.00 D) and of astigmatism (≤ 1.00 D)
* Neophyte contact lens wearer
* Be successfully fitted with spectacles or orthokeratology contact lenses
* Be able to achieve, through spherical refraction correction, a logMAR visual acuity of 0.8 or better in each eye
* Be willing and able to follow the subject instructions and to meet the protocol-specified schedule of follow-up visits
* White European ethnicity

Exclusion Criteria:

* Systemic or ocular disease affecting ocular health
* Use of any systemic or topical medications that could affect ocular physiology or contact lens performance
* Any lid or anterior segment abnormalities for which contact lens wear could be contraindicated
* CCLRU grade ≥ 2 for any given anterior segment ocular clinical signs
* Aphakic, amblyopic, and atopic individuals
* Refractive astigmatism ≥ ½ spherical refraction
* Previous contact lens wear

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — White European
Enrollment: 69 (Actual)
Dates: Start 2007-03-01 (Actual); Primary Completion 2010-03-01 (Actual); Study Completion 2010-03-01 (Actual)

PRIMARY OUTCOMES:
Axial length | Two years
  To compare axial length growth between white children with myopia wearing Menicon Z Night orthokeratology contact lenses and distance single-vision glasses. Measurements of axial length (in millimeters) were taken with the Zeiss IOLMaster (Carl Zeiss Jena GmbH, Jena, Germany). Three separate measurements of axial length were recorded per subject and per visit, and a mean obtained.

SECONDARY OUTCOMES:
Adverse events | Two years
  To compare the incidence of adverse events between white children with myopia wearing Menicon Z Night orthokeratology contact lenses and distance single-vision glasses. Adverse events were classified into serious, significant, or non-significant. Recurrences of the same adverse event(s) in the same or fellow eye at any of the subsequent study visits were classified as separate events; bilateral events will be counted as two separate events. The incidence of adverse events was calculated as a percentage of eyes per annum.
Patient-reported outcomes | Two years
  To compare vision-related quality-of-life measures between children wearing Menicon Z Night orthokeratology contact lenses and distance single-vision glasses. The pediatric refractive error profile survey was used to compare patient-reported outcomes in terms of the vision-specific quality of life between children in the Menicon Z Night and control groups. The survey consists of 26 statements scored from 1 (poor quality of life) to 5 (good quality of life), then scaled from 0 to 100 by subtracting 1 from the raw score of each question and multiplying by 25. The mean score of all items was calculated as the overall score. The survey includes 11 scales: overall vision, near vision, far distance vision, symptoms, appearance, satisfaction, activities, academics, handling, peer perception, and overall score.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Santodomingo-Rubido J, Villa-Collar C, Gilmartin B, Gutierrez-Ortega R. Myopia control with orthokeratology contact lenses in Spain: refractive and biometric changes. Invest Ophthalmol Vis Sci. 2012 Jul 31;53(8):5060-5. doi: 10.1167/iovs.11-8005. PMID 22729437
- [Result] Santodomingo-Rubido J, Villa-Collar C, Gilmartin B, Gutierrez-Ortega R. Orthokeratology vs. spectacles: adverse events and discontinuations. Optom Vis Sci. 2012 Aug;89(8):1133-9. doi: 10.1097/OPX.0b013e318263c5af. PMID 22773180
- [Result] Santodomingo-Rubido J, Villa-Collar C, Gilmartin B, Gutierrez-Ortega R. Myopia control with orthokeratology contact lenses in Spain: a comparison of vision-related quality-of-life measures between orthokeratology contact lenses and single-vision spectacles. Eye Contact Lens. 2013 Mar;39(2):153-7. doi: 10.1097/ICL.0b013e31827a0241. PMID 23392299